CLINICAL TRIAL: NCT04676529
Title: A Phase 1/2a Study to Evaluate Safety, Pharmacokinetic and Pharmacodynamic Dose Escalation and Expansion Study of PXS-5505 in Patients With Primary, Postpolycythemia Vera or Post-essential Thrombocythemia Myelofibrosis
Brief Title: Study to Evaluate Safety, Pharmacokinetic and Pharmacodynamic Dose Escalation and Expansion Study of PXS-5505 in Patients With Primary, Post-polycythemia Vera or Post-essential Thrombocythemia Myelofibrosis
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Syntara (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: PXS5505-MF-101
Record Dates: First submitted 2020-12-08; First posted 2020-12-21 (Actual); Last update posted 2025-08-24 (Actual); Status verified 2025-08

CONDITIONS: Myelofibrosis
Keywords: Thrombocythemia myelofibrosis; PXS-5505; Post polycythemia vera myelofibrosis
MeSH Terms: conditions — Primary Myelofibrosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- PXS-5505, Dose Level 1, Escalation Phase (Cohort A) (Experimental): Patients will receive PXS-5505 dose level 1, twice daily for a period of 4 weeks.
  Interventions: Drug: PXS-5505
- PXS-5505, Dose Level 2, Escalation Phase (Cohort B) (Experimental): Patients will receive PXS-5505 dose level 2, twice daily for a period of 4 weeks.
  Interventions: Drug: PXS-5505
- PXS-5505, Dose Level 3, Escalation Phase (Cohort C) (Experimental): Patients will receive PXS-5505 dose level 3, twice daily for a period of 4 weeks.
  Interventions: Drug: PXS-5505
- PXS-5505, Expansion Phase (Experimental): All patients will receive PXS-5505 at the selected twice daily dose for a period of 24 weeks, or until progressive disease, unacceptable toxicity, dose-limiting toxicity or withdrawal of consent.
  Interventions: Drug: PXS-5505
- PXS-5505, Add-on Phase (Experimental): Patients already receiving a stable dose of ruxolitinib for at least 12 weeks, will receive PXS-5505 (the dose used in the cohort expansion phase) on top of their ruxolitinib dose for up to 52 weeks or until progressive disease, unacceptable toxicity, dose-limiting toxicity, or withdrawal of consent.
  Interventions: Drug: PXS-5505

INTERVENTIONS:
Drug: PXS-5505 — PXS-5505 is a hard capsule (size 0) with the additional excipients mannitol and magnesium stearate.

SUMMARY:
This study will be an open-label phase 1/2a study to evaluate the safety and tolerability of PXS-5505 in patients with primary, postpolycythemia vera (PV) or post-essential thrombocythemia (ET) myelofibrosis.

DETAILED DESCRIPTION:
The study consists of three phases: a dose escalation phase, a cohort expansion phase, and an add-on phase.

The dose escalation phase will follow a 3+3 design with a starting dose of 100 mg twice daily, and a treatment duration of 4 weeks. Patients will be able to participate in more than one dose level.

During the cohort expansion phase, up to 24 patients will be treated at the dose determined appropriate based on safety, pharmacokinetic and pharmacodynamic results from the dose escalation phase, for a period of up to 6 months. Patients from the dose escalation phase will be able to participate in the cohort expansion phase.

In the add-on phase PXS-5505 will be given to patients, already receiving a stable dose of ruxolitinib, for a period of 12 months. Up to 15 patients will enrol in the add-on phase in order to obtain 12 patients with at least 1 month's exposure to PXS-5505 on top of ruxolitinib.

Note: The decision to include an add-on phase, where PXS-5505 is to be given on top of a stable ruxolitinib dose, was taken following a review of the data (safety, PK and PD) from the cohort expansion phase.

There will be no washout period between dose escalation and dose expansion cohorts.

ELIGIBILITY:
Inclusion Criteria:

* Have a pathologically confirmed established diagnosis of primary myelofibrosis or post-essential thrombocythemia/polycythemia vera myelofibrosis as per the World Health Organization 2016 diagnostic criteria (must include at least Grade 2 marrow fibrosis)
* Patients who are not eligible for stem cell transplantation
* a) Dose escalation / Cohort expansion phase only: Patients not currently on ruxolitinib or fedratinib (where available) treatment due to ineligibility, or previously treated patients who have been discontinued for at least 2 weeks prior to first dose of study drug due to any of the following criteria:

  * Ineligible: Platelets <50 x 10^9/L
  * Intolerant: Development of red blood cell transfusion dependence of at least two units/month for 2 months OR ≥Grade 3 adverse events of thrombocytopenia, anemia, hematoma, and/or hemorrhage while on treatment with ruxolitinib or fedratinib for at least 28 days
  * Refractory: < 10% spleen volume reduction by MRI or CT, or < 30% decrease from baseline in spleen volume by palpation after at least 3 months treatment with ruxolitinib or fedratinib
  * Relapsed: Regrowth to < 10% spleen volume reduction by MRI or CT, or < 30% decrease from baseline in spleen volume by palpation, following an initial response to ruxolitinib or fedratinib and after at least 3 months treatment
* b) Add-on phase only: Are being treated with ruxolitinib for at least 12 weeks prior to first administration of study treatment. The patient must be on a stable dose (no dose adjustments) of ruxolitinib for ≥ 8 weeks prior to study treatment and have not achieved complete remission (CR) by International Working Group (IWG) criteria.
* Have intermediate -2, or high-risk disease according to the International Working Group prognostic scoring system (DIPSS);
* a) Dose escalation / Cohort expansion phase only: Have symptomatic disease according to the MFSAF v4.0; Symptomatic disease is defined as a score of at least one in at least two items of the MFSAF v4.0;

  b) Add-on phase only: have a score of ≥ 10 on the MFSAF v4.0;
* Have symptomatic disease according to the MFSAF v4.0;
* Life expectancy of six months or greater;
* Must have adequate organ function as demonstrated by the following (within last 2 weeks):

  * Alanine aminotransferase and/or aspartate aminotransferase ≤ 2.5x upper limit of normal (ULN), or ≤ 4 x ULN (if upon judgment of the treating physician, it is believed to be due to extramedullary hematopoiesis [EMH] related to MF);
  * Direct bilirubin ≤ 1.5 x ULN; or ≤ 2 x ULN (if upon judgment of the treating physician, it is believed to be due to EMH related to MF);
  * Estimated glomerular filtration rate (eGFR) > 50 mL/min
* Eastern Cooperative Oncology Group performance status ≤ 2;
* Men must agree to using one medically approved contraceptive measure and have their partners agree to an additional barrier method of contraception for the duration of the study and for 90 days after the last administration of study drug; women of childbearing potential must use effective contraception
* Cohort Expansion and Add-on Phase only: A bone marrow biopsy must have been performed within 3 months prior to Day 1 treatment to establish the baseline fibrosis score or within 6 months of the re-initiation of treatment with PXS-5505 if subject participated in dose escalation phase of the trial

Exclusion Criteria:

* Greater than (>) 10% blasts in peripheral blood (determined within last two weeks);
* Prior splenectomy, or planning to undergo splenectomy, or splenic irradiation within 3 months prior to the first dose of study treatment
* Any serious medical condition or psychiatric illness that would prevent (as judged by the treating physician) the subject from signing the informed consent form or any condition, including the presence of laboratory abnormalities, which places the subject at unacceptable risk if he/she were to participate in the study or confounds the ability to interpret data from the study
* Known history of human immunodeficiency virus, active hepatitis C, or active hepatitis B
* History or presence of any form of cancer within the three years prior to enrolment, with the exception of excised basal cell or squamous cell carcinoma of the skin, or cervical carcinoma in situ or breast carcinoma in situ that has been excised or resected completely and is without evidence of local recurrence or metastasis
* Participation in an investigational drug or device trial within two weeks prior to study Day 1 or within five times the half-life of the investigational agent in the other clinical study, if known
* Use of any cytotoxic chemotherapeutic agents, including hydroxyurea, corticosteroids (prednisone ≤ 10 mg/day or corticosteroid equivalent is allowed), or immune modulators (e.g., thalidomide) within two weeks and interferon use within four weeks prior to study Day 1
* Symptomatic congestive heart failure (New York Heart Association Classification Class II), unstable angina, or unstable cardiac arrhythmia requiring medication
* Pregnancy
* History of surgery within two weeks prior to enrolment or anticipated surgery during the study period or two weeks post-study
* History of aneurysm
* Any other condition that might reduce the chance of obtaining data required by the protocol or that might compromise the ability to give truly informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2021-02-18 (Actual); Primary Completion 2025-07-09 (Actual); Study Completion 2025-07-09 (Actual)

PRIMARY OUTCOMES:
Number of subjects with serious and non-serious adverse events | Day 0 to follow-up visit (28 days -1 to +7days post-Tx discontinuation [dose escalation phase]; Day 0 to 28 days ± 3 days post-Tx discontinuation [cohort expansion phase]); Day 0 to follow-up visit (28 days ± 3 days post-Tx discontinuation [add-on phase]
  Safety and tolerability of PXS-5505 in patients with myelofibrosis will be assessed

SECONDARY OUTCOMES:
Maximum plasma concentration (C1hr=Cmax) | Day 0, week 1 and week 4 (dose escalation), and Day 0, week 4, 12 and 24 (cohort expansion and add-on phase), and week 52 during add-on phase only
  Pharmacokinetic parameters of PXS-5505 in patients with myelofibrosis will be assessed.
Minimum plasma concentration (Cmin) | Day 0, week 1 and week 4 (dose escalation), and Day 0, week 4, 12 and 24 (cohort expansion and add-on phase), and week 52 during add-on phase only
  Pharmacokinetic parameters of PXS-5505 in patients with myelofibrosis will be assessed.
Lysyl oxidase and lysyl oxidase-like 2 inhibition in plasma | Day 0, week 1 and week 4 dose escalation, and at week 0, 4, 12, 24 (cohort expansion and add-on phase), and week 52 during add-on phase only
  Pharmacodynamic parameters of PXS-5505 in patients with myelofibrosis will be assessed.
Change in bone marrow (BM) fibrosis | Day 0, Week 12 and Week 24 (cohort expansion and add-on phase), and week 52 during add-on phase only
  Change in bone marrow fibrosis will be assessed according to European Consensus on grading of bone marrow fibrosis
Response rate | At week 12 and week 24 (cohort expansion and add-on phase), weeks 38 and 52 during add-on phase only
  Response rates as defined by International Working Group (IWG)-Myeloproliferative Neoplasms Research and Treatment criteria in patients with myelofibrosis administered PXS-5505 will be determined.
Changes in spleen volume | Day 0, week 12, and week 24 (cohort expansion and add-on phase), weeks 38 and 52 during add-on phase only
  Changes in spleen volume, as measured by computed tomography (CT) or magnetic resonance imaging (MRI) scan, in patients with myelofibrosis administered PXS-5505 will be determined.
Changes in myelofibrosis related symptoms | Screening, week 12, and week 24 (cohort expansion and add-on phase), weeks 38 and 52 during add-on phase only
  Changes in myelofibrosis related symptoms based on Myelofibrosis-Symptom Assessment Form (MFSAF) v4.0 scores, in patients with myelofibrosis administered PXS-5505 will be determined. A higher score indicates worse symptoms.
Percentage of patients with hematological changes | Day 0, week 12, and 24 (cohort expansion and add-on phase), weeks 38 and 52 during add-on phase only
  Hematological changes will be determined

CONTACTS AND LOCATIONS:
Overall Officials: Jana Baskar, MBBS MMedSc MBA, Study Director — Syntara
Locations (23):
- United States (3):
  - Comprehensive Cancer Center (UAB CCC), Birmingham, Alabama
  - Novant Health Cancer Institute, Winston-Salem, North Carolina
  - The University of Texas MD Anderson Cancer Center, Houston, Texas
- Australia (5):
  - Liverpool Hospital, Liverpool, New South Wales
  - Ashford Cancer Centre Research, Adelaide, South Australia
  - St Vincent's Hospital Melbourne, Fitzroy, Victoria
  - One Clinical Research, Perth, Western Australia
  - The Perth Blood Institute, West Perth, Western Australia
- South Korea (10):
  - Inje University Busan Paik Hospital - Internal Medicine, Busan, Busan Gwang'yeogsi [Pusan-Kwan
  - Keimyung University Dongsan Hospital, Daegu, Daegu Gwang'yeogsi [Taegu-Kwangyokshi]
  - Gachon University Gil Hospital, Incheon, Incheon Gwang'yeogsi [Inch'n-K
  - National Cancer Center (Seoul Metro; northern), Gyeonggi-do
  - Seoul National University Hospital - Bundang, Gyeonggi-do
  - Seoul National University Hospital, Seoul
  - Severance Hospital, Yonsei University Health System- Haemat, Seoul
  - Asan Medical Centre, Seoul
  - Samsung Medical Center, Seoul
  - The Catholic University of Korea, Seoul St. Mary's Hospital, Seoul
- Taiwan (5):
  - Chang Gung Medical Foundation - ChiaYi Chang Gung Memorial Hospital - Hematology and Oncology, Chiayi City, Chiayi
  - Kaohsiung Medical University Chung-Ho Memorial Hospital, Kaohsiung City
  - China Medical University Hospital - Internal Medicine - Taichung, Taichung
  - National Cheng Kung University Hospital, Tainan
  - National Taiwan University Hospital - Hematology And Oncology, Taipei

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Vachhani P, Tan P, Watson AM, Wu SJ, Baker R, Cheung S, Lee SE, Chen CC, Chen TY, Hsiao HH, Lee JH, Masarova L, Tan SY, Baskar J, Charlton B, Findlay A, Hamprecht D, Jarolimek W, Leadbetter J, Miller J, Morgan K, Zahoor A, Hobbs G. A phase I/IIa trial of PXS-5505, a novel pan-lysyl oxidase inhibitor, in advanced myelofibrosis. Haematologica. 2025 Oct 1;110(10):2376-2387. doi: 10.3324/haematol.2024.287231. Epub 2025 Apr 17. PMID 40241543